CLINICAL TRIAL: NCT01166178
Title: A 1-year, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy of Zoledronic Acid 5 mg (Aclasta®) on Bone Mineral Density in Patients With Multiple Sclerosis Followed by a 1-year Open-label Treatment Phase
Brief Title: Zoledronic Acid in MS-patients With Osteoporosis
Acronym: EXALT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446HDE40; 2009-011888-37 (EudraCT Number)
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-10

CONDITIONS: Osteoporosis; Multiple Sclerosis
Keywords: Multiple Sclerosis; Osteoporosis; Zoledronic Acid
MeSH Terms: conditions — Osteoporosis; Multiple Sclerosis | interventions — Zoledronic Acid; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic Acid (Experimental): Participants received zoledronic acid infusion in addition to calcium and vitamin D
  Interventions: Drug: Zoledronic Acid; Dietary Supplement: Calcium and Vitamin D combination
- Placebo (Placebo Comparator): Participants received placebo to zoledronic acid infusion in addition to calcium and vitamin D
  Interventions: Drug: Placebo; Dietary Supplement: Calcium and Vitamin D combination

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid 5 mg once a year via intravenous infusion
  Arms: Zoledronic Acid
Drug: Placebo — Placebo to zoledronic acid once a year via intravenous infusion
  Arms: Placebo
Dietary Supplement: Calcium and Vitamin D combination — Calcium 500 mg and Vitamin D 400 IU combined tablet, taken orally twice a day

SUMMARY:
This study is designed to evaluate the efficacy and safety of zoledronic acid 5 mg intravenous (i.v.) relative to placebo in Multiple Sclerosis (MS) patients with osteoporosis and to support the optimal use of zoledronic acid for this indication. Primary objective is the change of Bone Mineral Density (BMD) at lumbar spine (L1-L4) and total hip region assessed by T-Score at month 12 relative to screening as measured by Dual X-ray Absorptiometry (DXA). This double-blind period will be followed by a 52-week open-label treatment phase to assess long-term efficacy and safety of zoledronic acid in these patients.

ELIGIBILITY:
Inclusion:

* Written informed consent to participate in the trial
* Definite diagnosis of Multiple Sclerosis (MS) as defined by 2005 revised McDonald criteria
* MS-subtype: Relapsing-remitting MS (RRMS), Secondary progressive MS (SPMS), Primary progressive MS (PPMS)
* Expanded Disability Status Scale (Kurtzke's scale; EDSS) score between 2.5 to 6.5 (including both)
* Bone mineral density (BMD) T-score of less or equal to -2.0 and more or equal to -4.0 at the lumbar spine (L1-L4 with at least 2 evaluable vertebrae) and/or total hip region and/or femoral neck in recent Dual X-Ray Absorptiometry (DXA)-scan (< or = 3 months)
* Sufficient ability to read, write and communicate comprehensibly and comply to study procedures
* No immunomodulatory treatment for MS within the last 30 days or stable and well tolerated therapy with any beta-interferon formulation, or glatirameracetate or fingolimod for at least 30 days immediately prior to baseline

Exclusion criteria:

* Contraindications against Calcium and Vitamin D and zoledronic acid according to the summary product characteristics
* More than one osteoporotic fracture
* Concomitant medication with influence on bone mineral density (eg. enzyme- inducing antiepileptics like Carbamazepin, Phenytoin, Phenobarbital, Primidon)
* Any neurological disorder other than MS which is known to affect bone mineral density (e.g. muscular dystrophy, severe paresis for other reasons than MS, degenerative nervous disorder, stroke)
* Women who are pregnant or breast feeding, or menstruating and capable of becoming pregnant.
* Baseline renal insufficiency
* 25-OH vitamin D level < 10 ng/ml at screening
* Serum calcium levels > 2.75 mmol/l (11.0 mg/dL) or < 2.00 mmol/L (8.0 mg/dL) at screening
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Germany (15):
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kassel
  - Novartis investigative site, Leipzig
  - Novartis Investigative Site, Leverkusen
  - Novartis investigative site, Ludwigshafen
  - Novartis investigative site, Magdeburg
  - Novartis investigative site, München
  - Novartis investigative site, Nümbrecht
  - Novartis investigative site, Oldenburg
  - Novartis Investigative Site, Siegen
  - Novartis investigative site, Stade

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 168 participants were planned to be randomized. 29 participants were randomized in a 2:1 ratio (zoledronic acid : placebo); no participants completed the study. One participant withdrew consent and the study was terminated.
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 21 | 8
Completed | 0 | 0
Not Completed | 21 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study was terminated | 20 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 21 | 8 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.0) | 56.0 (8.2) | 59.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density of the Lumbar Spine at 12 Months
Description: Change in bone mineral density (BMD) of the lumbar spine was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 12.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 12
Population: A total of 168 randomized participants were needed to have a power of 93% % to detect a significant difference in lumbar spine BMD. This study randomized 29 participants of the planned 168; hence, the planned analysis was not done.
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Bone Mineral Density of the Lumbar Spine at 6 Months
Description: Change in bone mineral density (BMD) of the lumbar spine was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 6.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 6
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Bone Mineral Density of the Femoral Neck at 6 Months
Description: Change in bone mineral density (BMD) of the femoral neck was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 6.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 6
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Bone Mineral Density of the Total Hip at 6 Months
Description: Change in bone mineral density (BMD) of the total hip was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 6. A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 6
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Bone Mineral Density of the Femoral Neck at 12 Months
Description: Change in bone mineral density (BMD) of the femoral neck was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 12.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 12
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Bone Mineral Density of the Lumbar Spine at 24 Months
Description: Change in bone mineral density (BMD) of the lumbar spine was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 24.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 24
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Change in Bone Mineral Density of the Total Hip Region at 12 Months
Description: Change in bone mineral density (BMD) of the total hip region was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 12.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 12
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Bone Mineral Density of the Total Hip Region at 24 Months
Description: Change in bone mineral density (BMD) of the total hip region was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 24.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 24
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Bone Mineral Density of the Femoral Neck at 24 Months
Description: Change in bone mineral density (BMD) of the femoral neck was measured using Dual X-ray Absorptiometry (DXA) at screening and at month 24.
  A DXA scanner is a device that uses x-ray beams to measure the amount of minerals in the bone.
Time Frame: Screening (day -21 to -1) and month 24
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Course of Disease in Multiple Sclerosis Patients
Description: The course of disease in Multiple Sclerosis (MS) patients was measured comparing results from the Expanded Disability Status Scale (EDSS) from screening and month 12. EDSS is a scale, ranging from 0 (normal) to 10 (death due to MS) for assessing neurologic impairment in MS. It is based on a weighting scheme of eight functional systems. The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel&Bladder, Cerebral and Other functions. EDSS was assessed by the treating neurologist.
Time Frame: Screening (day -21 to -1) and month 12
Population: as for outcome 1
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Adverse Events and Serious Adverse Events Comparison of Treatment Groups
Description: Adverse Events and Serious Adverse events are reported in the safety section.
Time Frame: 24 months
Population: A total of 168 randomized participants were needed to have a power of 93% % to detect a significant difference in lumbar spine BMD. This study randomized 29 participants of the planned 168; hence, the planned analysis was not done. The sample size was not powered for comparison between groups; however, all AEs are reported in the safety section.
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/8
Other Adverse Events (participants affected / at risk) | 16/21 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid (N=21) | Placebo (N=8)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=21) | Placebo (N=8)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1
FATIGUE (General disorders) | 2 | 0
GAIT DISTURBANCE (General disorders) | 1 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 7 | 1
PYREXIA (General disorders) | 1 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 2
DIZZINESS (Nervous system disorders) | 1 | 2
HEADACHE (Nervous system disorders) | 7 | 2
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Study termination due to small number of participants recruited lead to lack of power for analysis of all outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.